CLINICAL TRIAL: NCT05384366
Title: To Study the Factors Affecting Treatment Responses in Patients With Uterine Cervical Carcinoma Undergoing Neoadjuvant Chemotherapy
Brief Title: Neoadjuvant Chemotherapy in Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Banaras Hindu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoCx
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cervix Cancer; Cervical Cancer; Cancer of the Uterine Cervix
Keywords: cancer; cervix; neoadjuvant chemotherapy; predictors
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — Neoadjuvant Therapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Patients with locally advanced carcinoma of the uterine cervix were recruited for assessment of clinical and pathological therapeutic response. Multivariate analysis was conducted to predict the independent predictors of response
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy (Other): Patients receiving neoadjuvant paclitaxel 175mg/m2 and carboplatin (AUC5) at three weekly interval by intravenous route
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — doublet of taxane and carboplatin
  Other Names: Paclitaxel and Carboplatin

SUMMARY:
Cervical cancer represents the second commonest cancer in women worldwide, with 500,000 new cases and 300,000 deaths reported yearly. Among cervical cancer cases, 80% occur in developing countries and about 70% are identified as advanced cancer. According to the International Federation of Gynecology and Obstetrics (FIGO) staging system, a locally advanced cervical cancer includes stage IB2 to IIB.

Treatment modalities include radical surgery with or without adjuvant radiotherapy (RT), Neoadjuvant Chemotherapy (NAC) plus radical hysterectomy with or without adjuvant RT, and concomitant chemo radiation. Currently, platinum based concurrent chemoradiotherapy is the gold standard for locally advanced cervical carcinoma.

Neoadjuvant chemotherapy has many advantages: decreasing tumor size making surgery easier with improved rate of complete resection, decreased pelvic recurrence rate significantly, decreasing rate of parametrial invasion and lymph node metastasis, better brachytherapy distribution, minimal radiation toxicity, and 15% absolute increase of 5-year survival.

This study will evaluate various factors i.e. patient related (Age, Menopausal status, HPV, HIV, Comorbidities), Tumor related pathological stages (TNM), grade, lymphovascular perineural invasion, lymph nodes, extranodal extension, tumor margins including radial margin, type of tumor i.e. Adeno vs squamous, mutation profile and Treatment related factors (type of NAC, duration of NAC, no of cycles of NAC).

DETAILED DESCRIPTION:
This is a single group prospective study to evaluate factors affecting treatment responses in uterine cervical carcinoma. All patients who will be receiving NAC followed by surgery will be included and assessed for various defined factors influencing response. Responses will be assessed by RECIST 1.1 criteria.

1. All patients of cervical growth will be evaluated. Initial clinical evaluation, biopsy and if positive, HPV DNA status will be done. On confirmation of malignancy further staging will be done by FIGO Classification. Imaging will include contrast enhanced computed tomography (CECT) abdomen or Magnetic resonance imaging (MRI) pelvis and ultrasound (USG) abdomen. Routine blood investigations, chest X-ray (CXR) and Electrocardiography (ECG) will be done.
2. In recruited patients, 3 cycles of NAC consisting of Paclitaxel (175 mg/m2) and Carboplatin (AUC5) at 21 day intervals were given.
3. Adverse reactions if any were recorded as WHO toxicity grades.
4. Evaluation of response was done after end of 2nd cycle of chemotherapy with clinical examination and Imaging (CT/MRI) by RECIST 1.1 criteria.
5. Response was divided into two groups- 1) Complete/ Partial response 2) Poor response/ Stable disease/ Progressive disease. Patients with Poor response/ stable disease/ progressive disease will undergo concurrent chemoradiation (CCRT) while patients with partial/complete response will undergo Wertheim's hysterectomy.
6. After surgery Pathological evaluation will include T, N, M, histological type, Lymphovascular invasion (LVI), Perineural invasion (PNI), Depth of Tumor Invasion, Extra nodal extension (ENE), Grade, (next generation sequencing (NGS)- Mutation Analysis.
7. Post operative external pelvic irradiation was given according to Sedlis criteria in node negative, margin negative, parametria negative cases.
8. Follow up Evaluation was done at 1, 3 & 6 months by clinical examination, Biopsy for any recurrence and Imaging (CECT or MRI pelvis) at 6 months. Follow up was continued every 3 months thereof.

ELIGIBILITY:
Inclusion Criteria:

* • All patients receiving NACT followed by Surgery/RT and willing to give consent will be included in study

  * FIGO Stage Ib/ IIa/ IIb
  * Age more than 18 yrs

Exclusion Criteria:

* • FIGO Stage Ia/ III/ IV

  * Patients who received treatment earlier
  * Pregnant/ lactating women
  * Second primary cancer

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The disease occurs only in females
Enrollment: 33 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 21 days after completion of third cycles
  Response to intervention by RACIST criteria 1.1
Pathological response | 6 months
  Pathological response after evaluation of surgical specimen and pathological staging

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, MS, PhD, Principal Investigator — Banaras Hindu University
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: on request

REFERENCES:
- [Background] Rose PG. Combined-modality therapy of locally advanced cervical cancer. J Clin Oncol. 2003 May 15;21(10 Suppl):211s-217s. doi: 10.1200/JCO.2003.01.222. PMID 12743137
- [Background] Katsumata N, Yoshikawa H, Kobayashi H, Saito T, Kuzuya K, Nakanishi T, Yasugi T, Yaegashi N, Yokota H, Kodama S, Mizunoe T, Hiura M, Kasamatsu T, Shibata T, Kamura T; Japan Clinical Oncology Group. Phase III randomised controlled trial of neoadjuvant chemotherapy plus radical surgery vs radical surgery alone for stages IB2, IIA2, and IIB cervical cancer: a Japan Clinical Oncology Group trial (JCOG 0102). Br J Cancer. 2013 May 28;108(10):1957-63. doi: 10.1038/bjc.2013.179. Epub 2013 May 2. PMID 23640393
- [Background] Singh U, Ahirwar N, Rani AK, Singh N, Sankhwar P, Qureshi S. The efficacy and safety of neoadjuvant chemotherapy in treatment of locally advanced carcinoma cervix. J Obstet Gynaecol India. 2013 Aug;63(4):273-8. doi: 10.1007/s13224-012-0342-6. Epub 2013 Mar 12. PMID 24431655
- [Background] Osman M. The role of neoadjuvant chemotherapy in the management of locally advanced cervix cancer: a systematic review. Oncol Rev. 2014 Sep 23;8(2):250. doi: 10.4081/oncol.2014.250. eCollection 2014 Sep 23. PMID 25992238
- [Background] Sardi JE, Giaroli A, Sananes C, Ferreira M, Soderini A, Bermudez A, Snaidas L, Vighi S, Gomez Rueda N, di Paola G. Long-term follow-up of the first randomized trial using neoadjuvant chemotherapy in stage Ib squamous carcinoma of the cervix: the final results. Gynecol Oncol. 1997 Oct;67(1):61-9. doi: 10.1006/gyno.1997.4812. PMID 9345358
- [Background] Takatori E, Shoji T, Omi H, Kagabu M, Miura F, Takeuchi S, Kumagai S, Yoshizaki A, Sato A, Sugiyama T. Analysis of prognostic factors for patients with bulky squamous cell carcinoma of the uterine cervix who underwent neoadjuvant chemotherapy followed by radical hysterectomy. Int J Clin Oncol. 2015 Apr;20(2):345-50. doi: 10.1007/s10147-014-0702-6. Epub 2014 May 14. PMID 24825458
- [Background] Koensgen D, Sehouli J, Belau A, Weiss M, Stope MB, Grokopf V, Eichbaum M, Ledwon P, Lichtenegger W, Zygmunt M, Kohler G, Mustea A. Clinical Outcome of Neoadjuvant Radiochemotherapy in Locally Advanced Cervical Cancer: Results of an Open Prospective, Multicenter Phase 2 Study of the North-Eastern German Society of Gynecological Oncology. Int J Gynecol Cancer. 2017 Mar;27(3):500-506. doi: 10.1097/IGC.0000000000000894. PMID 28187089
- [Background] Di Donato V, Schiavi MC, Ruscito I, Visentin VS, Palaia I, Marchetti C, Fischetti M, Monti M, Muzii L, Benedetti Panici P. Effects of Neoadjuvant Chemotherapy Plus Radical Surgery as Front Line Treatment Strategy in Patients Affected by FIGO Stage III Cervical Cancer. Ann Surg Oncol. 2016 Dec;23(Suppl 5):841-849. doi: 10.1245/s10434-016-5597-1. Epub 2016 Sep 27. PMID 27678502